CLINICAL TRIAL: NCT06227793
Title: Pragmatic Clinical Trial to Assess the Effectiveness of Pharmaceutical Intervention in Patients With Uncontrolled Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 20230013
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): With health education
  Interventions: Behavioral: pharmaceutical intervention
- control (No Intervention): Without health education

INTERVENTIONS:
Behavioral: pharmaceutical intervention — Individuals randomized to the intervention group will undergo monthly pharmaceutical consultations for health education, initiated after randomization. There will be three in-person consultations, starting in month 1 with monthly spacing, scheduled by the pharmacist in the office, except for the first consultation, which will be scheduled by the pharmacist over the phone after randomization. These consultations will be part of the intervention study's educational process and will take place between the initial and final assessments. The educational process scripts for each consultation include a pharmaceutical follow-up form and an inhalation technique assessment form. Once the consultation is completed, the patient will also receive, via WhatsApp and/or email according to their preference, an educational video demonstrating the step-by-step inhalation technique based on their prescribed treatment.
  Arms: intervention

SUMMARY:
The aim of this study is to evaluate the effectiveness of pharmaceutical intervention in controlling asthma in patients diagnosed with uncontrolled asthma. This is a pragmatic clinical trial composed of two groups - intervention (pharmaceutical monitoring) and control (without pharmaceutical monitoring). The study population will consist of patients with uncontrolled asthma, seen at the asthma outpatient clinic of the Hospital de Clínicas de Porto Alegre. Patients who agree to participate in the study will be randomized to the control group (managed by the specialized outpatient medical team) and the intervention group (in addition to management by the specialized medical team, they will be referred for pharmaceutical monitoring at the Clinical Research Center of the Hospital de Clínicas de Porto Alegre). The primary outcome of the study will be the proportion of patients with uncontrolled asthma who achieve an ACT > 20 after a systematic educational intervention, guided by a pharmaceutical professional, compared to a group that does not receive this type of intervention.

DETAILED DESCRIPTION:
Asthma is a heterogeneous disease, typically characterized by chronic inflammation of the airways. Uncontrolled asthma is a condition that can directly impact patients' quality of life and be associated with non-adherence to treatment and errors in inhalation technique. It is known that pharmaceutical monitoring contributes positively to asthma control. Thus, the aim of this study is to evaluate the effectiveness of pharmaceutical intervention in controlling asthma in patients diagnosed with uncontrolled asthma. This is a pragmatic clinical trial composed of two groups - intervention (pharmaceutical monitoring) and control (without pharmaceutical monitoring). The study population will consist of patients with uncontrolled asthma, seen at the asthma outpatient clinic of the Hospital de Clínicas de Porto Alegre. Patients who agree to participate in the study will be randomized to the control group (managed by the specialized outpatient medical team) and the intervention group (in addition to management by the specialized medical team, they will be referred for pharmaceutical monitoring at the Clinical Research Center of the Hospital de Clínicas de Porto Alegre). For both groups, the Asthma Control Test (ACT), the standardized Asthma Quality of Life Questionnaire (AQLQ(S)), and treatment adherence questionnaire will be administered by phone at the beginning of month 1 and at the end of month 3, by a blinded researcher in the study. The primary outcome of the study will be the proportion of patients with uncontrolled asthma who achieve an ACT > 20 after a systematic educational intervention, guided by a pharmaceutical professional, compared to a group that does not receive this type of intervention. To achieve this, a sample size of 50 individuals (25 for each group) was calculated to test for a difference between the percentages of controlled asthma (ACT > 20) at the end of 3 months between the Pharmaceutical Intervention and Control groups. With an additional 30% for possible losses and refusals, this number should be 56. The calculation considered a power of 80%, a significance level of 5%, and percentages of 50% and 10%, respectively. This study is expected to generate scientific evidence on the effectiveness of pharmaceutical intervention in asthma control and guide public policies within the Unified Health System (SUS).

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 70 years.
* Previous diagnosis of asthma according to clinical and pulmonary functional criteria, established in national and international guidelines.
* Present uncontrolled asthma as assessed by the ACT (score below 20 points) (32).
* Be undergoing outpatient treatment at the Pulmonology Service of HCPA for at least 6 months and have had at least 2 prior consultations.
* Reside in Porto Alegre or in the metropolitan region of Porto Alegre.
* Smoking index less than 10 pack-years (number of cigarettes smoked per day / 20 cigarettes x number of years of smoking).

Exclusion Criteria:

* Pregnant patients
* Chronic neurological or psychiatric diseases that prevent the execution of study procedures
* Pulmonary comorbidities such as chronic obstructive pulmonary disease, diffuse bronchiectasis, extensive sequelae of tuberculosis, diffuse pulmonary fibrosis.
* Lung neoplasms or from other sites.
* Incapacitating cardiovascular diseases
* Patients without access to WhatsApp.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Asthma control | 3 years
  The degree of asthma control will be determined according to the Asthma Control Test (ACT). The questionnaire score ranges from 5 to 25 (higher scores indicate better control), with a score of 25 points expressing the best possible control. Scores from 20 to 25 are classified as controlled; 16-19 as not well controlled; and 5-15 as very poorly controlled asthma. The ACT consists of four questions about symptoms/relief and self-assessment of control by the patient. A clinically important minimum difference of 3 points is considered.

SECONDARY OUTCOMES:
Degree of adherence to treatment | 3 years
  Treatment adherence will be measured through self-reported adherence, using a questionnaire employed in a study involving asthmatic patients as a reference. The adherence score will be defined as a score above 5 points or below 5 points. High adherence will be indicated when the reported use of devices containing corticosteroids is 5 or more times per week, while low adherence will be considered when it is less than 5 times per week.
Asthma Quality of Life Questionnaire | 3 years
  The quality of life will be assessed using The Asthma Quality of Life Questionnaire (AQLQ). The overall score of the questionnaire is the arithmetic mean of all items, with a minimum score of 1 and a maximum of 7 points. Higher scores would indicate better quality of life in relation to asthma.
Lung function (spirometry) | 3 years
  The spirometry used for the diagnosis of asthma will be obtained through a review of the patient's medical records or by query. The baseline spirometry for the study will be the one conducted during the routine medical consultation, also obtained through a review of medical records or by query. The study will include a spirometry test at the end of the 3 months, after the pharmaceutical interventions, to be requested by the research team. Spirometry tests are routinely performed in the Pulmonary Physiology Unit of the Pneumology Service at HCPA.
  Pneumologia do HCPA.
Rates of exacerbations requiring oral corticosteroid use | 3 years
  Clinical and demographic data will be recorded upon request through queries. For those that cannot be collected through queries, the information will be obtained directly from the medical records or gathered during the initial evaluation.
Emergency room visits for asthma | 3 years
  Clinical and demographic data will be recorded upon request through queries. For those that cannot be collected through queries, the information will be obtained directly from the medical records or gathered during the initial evaluation.
Hospital admissions due to asthma | 3 years
  Clinical and demographic data will be recorded upon request through queries. For those that cannot be collected through queries, the information will be obtained directly from the medical records or gathered during the initial evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Dalcin, Principal Investigator — Hospital Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No